CLINICAL TRIAL: NCT01265641
Title: A Single-centre, Double-blind, Double-dummy, Randomised, Placebo Controlled, Four-period Crossover Study in Healthy Male Volunteers, to Assess the Effect on QT/QTc Interval of Single Oral Doses of AZD1981 (200 mg and 2000 mg) Using Moxifloxacin (Avelox®) as a Positive Control
Brief Title: To Investigate the Effects of AZD1981 on the QT Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Christer Hultquist / MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D9830C00011; 2010-023338-22
Record Dates: First submitted 2010-12-17; First posted 2010-12-23 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — AZD1981; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: AZD1981, 2000mg
- 2 (Experimental)
  Interventions: Drug: AZD1981, 200mg
- 3 (Experimental)
  Interventions: Drug: Moxifloxacin, 400mg
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1981, 2000mg — Single oral dose, tablets
  Arms: 1
Drug: AZD1981, 200mg — Single oral dose, tablets
  Arms: 2
Drug: Moxifloxacin, 400mg — Single oral dose, capsule
  Arms: 3
Drug: Placebo — Single oral dose, tablets
  Arms: 4

SUMMARY:
The purpose of this research study is to evaluate the effect of AZD1981 on the electrical activity of the heart, in particular when the heart muscle is relaxed during a heart beat cycle. The effect of AZD1981 will be compared to a licensed antibiotic (moxifloxacin) which is well known to affect the electrical activity of the heart, but this effect is known to be at levels that are safe at the dose used in this study. The investigators will also compare the effects of AZD1981 with a "dummy drug" (placebo). The investigators will also be evaluating how safe and well tolerated AZD1981 is and how much AZD1981 enters the blood circulation by collecting blood during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 55 years (inclusive)
* Subjects must be willing to use barrier methods of contraception during study and for 3 months after last dosing.
* Be a non-smoker or ex-smoker who has stopped smoking for >6 months

Exclusion Criteria:

* Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment)
* History of additional risk factors for Torsade de Pointes (eg, heart failure, hypokalemia, personal or family history of arrhythmia or long QT syndrome)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of a single supra maximal therapeutic dose of AZD1981on QT interval - QTcF | dECG and telemetry measurements taken pre-dose and up to and including 48 hours post dose

SECONDARY OUTCOMES:
To evaluate the effect of a therapeutic dose of AZD1981on QT interval -QTcF | dECG and telemetry measurements taken pre-dose and up to and including 48 hours post dose
To evaluate the effect of AZD1981 on additional electrocardiogram variables - QTcB -RR PR QRS. | dECG and telemetry measurements taken pre-dose and up to and including 48 hours post dose
To evaluate the safety and tolerability of single doses of AZD1981 -frequency of adverse events - laboratory safety assessments - vital signs - physical examination - ECG. | Adverse events recorded at all four residential visits (one week washout between visits) and at follow up (7-10 days following last residential visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Researche Site, London, UK, United Kingdom